CLINICAL TRIAL: NCT04724941
Title: Prodromal Alpha-Synuclein Screening in Parkinson's Disease Study
Acronym: PASS-PD
Status: Recruiting | Type: Observational
Sponsor: University Hospital Schleswig-Holstein (Other)
Collaborators: UCB Biopharma SRL (Industry); University of Kiel (Other)
Responsible Party: Principal Investigator, Eva Schaeffer, Dr. Eva Schaeffer, Department for Neurology, University Hospital Schleswig-Holstein
Other Study IDs: PASS_PD_D440/2
Record Dates: First submitted 2021-01-21; First posted 2021-01-26 (Actual); Last update posted 2025-09-22 (Actual); Status verified 2025-09

CONDITIONS: Parkinson Disease
Keywords: Prodromal; Alpha-Synuclein; Risk disclosure
MeSH Terms: conditions — Parkinson Disease; Parkinson Disease 4, Autosomal Dominant Lewy Body

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- REM behavior disorder +: Individuals with REM Sleep Behavior Disorder:
  All individuals will be included in a prospective, longitudinal observational study, including an annual investigation at the Department for Neurology (detailed anamnesis, neurological examination, motor assessment). Blood sampling will be performed every six months, non-motor symptoms will be assessed every three months using online surveys. All individuals can participate in an optional substudy including lumbar punctures every two years.
  Interventions: Other: No intervention
- REM behavior disorder -: Individuals without REM Sleep Behavior Disorder with increased risk for PD:
  All individuals will be included in a prospective, longitudinal observational study, including an annual investigation at the Department for Neurology (detailed anamnesis, neurological examination, motor assessment). Blood sampling will be performed every six months, non-motor symptoms will be assessed every three months using online surveys. All individuals can participate in an optional substudy including lumbar punctures every two years.
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — No intervention

SUMMARY:
The PASS-PD study is set out to screen individuals from the general population with an increased risk for the development of Parkinson's Disease (PD) and to investigate this highly enriched cohort longitudinally for five year. A special focus is placed on implementation of ethical standards for early risk disclosure in PD.

DETAILED DESCRIPTION:
The PASS-PP Study is designed to combine the latest developments in clinical and biomarker research to

1. understand the distribution of risk profiles for PD in the general population, especially regarding non-motor symptoms
2. identify subjects with a likelihood of developing PD
3. follow individuals with a high likelihood/risk to develop PD in the future (compared to individuals with low risk and) in a prospective study
4. understand the potential of biological markers to increase prediction of progression/conversion
5. identify subtypes of PD patients, by providing a detailed clinical phenotyping with a main focus on non-motor symptoms cluster
6. provide a framework of ethical handling of early risk disclosure in PD

ELIGIBILITY:
Inclusion Criteria:

* Age between 50 and 99

Exclusion Criteria:

* Presence of clinical PD at the time of study inclusion
* Other significant neurologic diseases affecting the central nervous system (e.g. Multiple sclerosis)
* other significant diseases e.g. orthopaedic diseases affecting quantitative motor assessment
* in case of participation in the lumbal puncture substudy: contraindications for the performance of lumbal puncture (bleeding tendency, intake of anticoagulants)

Ages: 50 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: General population
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2021-06-01 (Actual); Primary Completion 2027-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Risk marker profile | Analysis after three years.
  Extend and progression of risk marker profile

SECONDARY OUTCOMES:
Non-motor and motor symptoms | Analysis after three years
  Development and progression of non-motor and motor symptoms

CONTACTS AND LOCATIONS:
Overall Officials: Daniela Berg, Prof.Dr., Principal Investigator — Department for Neurology, University of Kiel
Locations (1):
- Department for Neurology, University of Kiel, Kiel, Germany

IPD SHARING:
Plan to Share IPD: Undecided
After successful analysis and publication of data the clinical data can be shared upon request.